CLINICAL TRIAL: NCT00201045
Title: Collaborative Management of Hypertension
Brief Title: Team Management of High Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Barry L. Carter, The University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 271; R01HL069801 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2007-12

CONDITIONS: Hypertension
Keywords: Hypertension management; Pharmacist management; Physician pharmacist collaboration; Blood pressure control
MeSH Terms: conditions — Hypertension | interventions — Physicians

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Intervention patients receive care from a clinical pharmacist to improve blood pressure.
  Interventions: Other: Physician/Pharmacist Collaborative Teams
- Control (No Intervention): Control patients receive usual care and do not have a clinical pharmacist included in their care.

INTERVENTIONS:
Other: Physician/Pharmacist Collaborative Teams — The patient's physician collaborates with a clinical pharmacist to improve management of hypertension
  Arms: Intervention

SUMMARY:
The purpose of this study is to test whether blood pressure control can be improved by physician education and feedback provided through the development of physician/pharmacist collaborative teams.

DETAILED DESCRIPTION:
BACKGROUND:

The Healthy People 2010 target calls for controlled BP in 50% of the 50 million Americans with hypertension. BP is currently controlled in only 27% of the population. These population figures are in contrast to data from clinical trials (efficacy) in which BP has been controlled in 70 to 80% of study participants. Poor BP control exists in spite of six sets of guidelines generated over the last 30 years in the United States. While there are many causes for poor control, several studies have found that physicians are frequently satisfied with uncontrolled BPs. Numerous strategies exist to assist physicians with achieving better BP control, but a consistent, effective approach to solving the problem has not been found.

DESIGN NARRATIVE:

The objective of this study is to test whether BP control can be improved by physician education and feedback provided through the development of physician/pharmacist collaborative teams. The rationale for this proposal is generated from studies demonstrating that physician knowledge, quality of prescribing, and attainment of treatment goals can be improved when physicians collaborate with clinical pharmacists. Previous studies have suffered from insufficient sample size and controls and did not include a structured intervention. This study will address these gaps in knowledge by conducting a randomized, prospective study in 5 clinics (2 intervention and 3 control) with 27 physicians who care for 180 patients with uncontrolled BP. The structured intervention will involve clinical pharmacists who evaluate BP therapy and treatment strategies and make specific recommendations to the physician. Patients will be seen at baseline and at 2, 4, 6, 8, and 9 months, at which time random zero BP measurements will be performed. The specific aims of this study are (1) to determine if better BP control can be achieved by the use of physician/pharmacist teams that utilize physician education and feedback when compared to usual care, (2) to determine if improvements in BP control are related to an increase in physician knowledge of and adherence to BP guidelines when they are involved in physician/pharmacist teams, and (3) to determine if changes in BP control are associated with the level and scope of the physician/pharmacist relationships. This model utilizes an innovative system approach to improve BP control. This intervention has the potential to achieve marked improvements in BP control. This model could become one additional strategy to help achieve the BP goals for Healthy People 2010.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, age 21-85
* Taking 0-3 antihypertensive medications with no changes in regimen or dose within the past 4 weeks
* Non-diabetic with clinic BP 145-179 / 95-109 or diabetic with BP greater than 135/85

Exclusion Criteria:

* Previous 24 hour BP monitoring consult service within the past 6 months
* Stage 3 hypertension greater than 180/110
* Recent MI or stroke within the past 6 months
* Class III or IV congestive heart failure
* Unstable angina
* Uncontrolled atrial fibrillation
* Serious renal disease (serum creatinine greater than 3.5)
* Serious hepatic disease (total bilirubin greater than 3.0)
* Pregnancy
* Poor prognosis with less than a 3 year life expectancy

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2003-07; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Blood pressure control | Measured by zero blood pressure measurements at baseline and 2, 4, 6, 8, and 9 months

SECONDARY OUTCOMES:
Mean number of antihypertensives | Measured when each patient completed the study.
Side effect score | Measured when each patient completed the study.
Physician knowledge | Measured at the beginning and at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Barry L. Carter, Study Chair — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Background] Carter BL, Hartz A, Bergus G, Dawson JD, Doucette WR, Stewart JJ, Xu Y. Relationship between physician knowledge of hypertension and blood pressure control. J Clin Hypertens (Greenwich). 2006 Jul;8(7):481-6. doi: 10.1111/j.1524-6175.2006.05601.x. PMID 16849901
- [Background] Carter BL. Antihypertensive prescribing: do we have reason to celebrate? Hypertension. 2006 Nov;48(5):816-7. doi: 10.1161/01.HYP.0000240978.77934.3a. Epub 2006 Sep 18. No abstract available. PMID 16982966
- [Background] Carter BL, Sica DA. Strategies to improve the cardiovascular risk profile of thiazide-type diuretics as used in the management of hypertension. Expert Opin Drug Saf. 2007 Sep;6(5):583-94. doi: 10.1517/14740338.6.5.583. PMID 17877445
- [Background] Carter BL, Rogers M, Daly J, Zheng S, James PA. The potency of team-based care interventions for hypertension: a meta-analysis. Arch Intern Med. 2009 Oct 26;169(19):1748-55. doi: 10.1001/archinternmed.2009.316. PMID 19858431
- [Result] Carter BL, Bergus GR, Dawson JD, Farris KB, Doucette WR, Chrischilles EA, Hartz AJ. A cluster randomized trial to evaluate physician/pharmacist collaboration to improve blood pressure control. J Clin Hypertens (Greenwich). 2008 Apr;10(4):260-71. doi: 10.1111/j.1751-7176.2008.07434.x. PMID 18401223
- [Derived] Weber CA, Ernst ME, Sezate GS, Zheng S, Carter BL. Pharmacist-physician comanagement of hypertension and reduction in 24-hour ambulatory blood pressures. Arch Intern Med. 2010 Oct 11;170(18):1634-9. doi: 10.1001/archinternmed.2010.349. PMID 20937921